CLINICAL TRIAL: NCT01578226
Title: Role of Procalcitonin (PCT) for the Diagnosis of Sepsis in Ascitic Cirrhotic Patients
Brief Title: Procalcitonin in Cirrhotic Patients at High Risk for Sepsis
Status: Completed | Type: Observational
Sponsor: Prof. Facchinetti Fabio (Other)
Responsible Party: Sponsor-Investigator, Prof. Facchinetti Fabio, PRS Admin, University of Modena and Reggio Emilia
Organization: University of Modena and Reggio Emilia (Other)
Other Study IDs: PCTCIRR
Record Dates: First submitted 2012-04-13; First posted 2012-04-16 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Cirrhosis; Ascites; Sepsis
Keywords: Cirrhosis; Ascites; Decompensation; Bacterial infection; Sepsis; Procalcitonin; PCT
MeSH Terms: conditions — Fibrosis; Ascites; Sepsis; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Decompensated cirrhotic patients: Cirrhotic patients presenting with clinically detectable ascites (Grade 2 o Grade 3)

SUMMARY:
Infections are frequent life-threatening events in patients with cirrhosis, occurring at least in 35% of hospitalized patients and accounting for 20% of inpatients death. Among cirrhotics, ascitic patients have the highest risk of death for sepsis. At the admission, no clear-cut clinical and biochemical features are helpful in diagnosing and prognostically stratifying those patients with sepsis. Procalcitonin (PCT)is a breakthrough marker presenting high sensibility and specificity in diagnosing bacterial infections in different clinical settings. The purpose of this study is to evaluate PCT as a diagnostic and prognostic tool for sepsis in hospitalized cirrhotic patients with ascitic decompensation.

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis regardless of aetiology
* clinically relevant ascitic decompensation at time of hospital admission

Exclusion Criteria:

* high haematic ascites
* ongoing antimicrobial therapy or stopped less than 7 days before admission
* last hospital discharge within 7 days
* surgery or trauma within 30 days from enrolment
* hepatocellular carcinoma out of Milan criteria
* extra hepatic malignancies
* immunodeficiency syndrome
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ascitic cirrhotic patients admitted to our third level Liver Unit.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Schepis, MD, Principal Investigator — University of Modena and Reggio Emilia
Locations (1):
- Gastroenterology Unit - University Hospital of Modena, Modena, Italy